CLINICAL TRIAL: NCT00418418
Title: Combined CABG and Stem-Cell Transplantation for Heart Failure
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Helsinki (Other)
Responsible Party: Reijo Haapiainen, Helsinki University Hospital
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TYH 6220
Record Dates: First submitted 2007-01-03; First posted 2007-01-04 (Estimated); Last update posted 2008-08-19 (Estimated); Status verified 2008-08

CONDITIONS: Heart Failure; Myocardial Infarction; Coronary Artery Disease
Keywords: Cell transplantation; Heart failure; Clinical trials
MeSH Terms: conditions — Heart Failure; Myocardial Infarction; Coronary Artery Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Active Comparator): Patient group receiving the stem cell injections during the CABG
  Interventions: Procedure: Coronary bypass operation; Procedure: Bone marrow aspiration (crista iliaca); Biological: Intramyocardial mesenchymal stem cell transplantation
- B (Placebo Comparator): The patient group receiving autologous serum injections during the CAGB operation
  Interventions: Procedure: Coronary bypass operation; Procedure: Bone marrow aspiration (crista iliaca); Biological: Intramyocardial injection of autologous serum

INTERVENTIONS:
Procedure: Coronary bypass operation — Coronary bypass operation is performed via sternotomy during cardiac arrest.
  Other Names: CABG
Procedure: Bone marrow aspiration (crista iliaca) — The bone marrow is aspirated from the iliac crest (100ml). During the operation the aspirate is transported to the stem cell laboratory, where the sample is centrifugated through Ficoll(Registered Trademark).
  Other Names: Stem cell harvest
Biological: Intramyocardial mesenchymal stem cell transplantation — During the cardiac arrest, stem cells are directly injected to myocardium. The amount of the cells varies individually (5-1000 x 10e6 cells), the cells are diluted in autologous serum (5 ml)
  Other Names: Stem cell therapy
  Arms: A
Biological: Intramyocardial injection of autologous serum — Intramyocardial injection of autologous serum is injected during cardiac arrest
  Other Names: Stem cell control therapy
  Arms: B

SUMMARY:
This is a prospective double blind trial of intraoperative transmyocardial bone marrow-derived mesenchymal cell transplantation vs placebo in patients with low left ventricular ejection fraction scheduled to coronary bypass operation.

DETAILED DESCRIPTION:
The prevalence of symptomatic heart failure in general population is up to 2% and the prevalence increases rapidly with age. Half of the patients with symptomatic heart failure will die within 4 years of diagnosis.The purpose of this study is to examine the effect of bone marrow-derived stem cell transplantation in left ventricular ejection fraction.

Consecutive patients with systolic heart failure (n=60), with ischemic coronary heart disease, scheduled to by-pass-operation (CABG) will be collected from cardiovascular laboratory and outpatient clinic of Helsinki University Central Hospital. Patients should have heart failure with ejection fraction between 15 to 45%. Randomly patients are selected to receive a stem cell transplantation with best possible heart failure medication, or without cell transplantation. In this study, 30 patients are receiving bone marrow transplantation, and 30 patients are serving as a control population. All patients will receive CABG.The study will be carried out with randomized, double blind techniques for one year. Randomization (in blocks) will be based on a table of random numbers.Bone marrow and patients own serum will be blinded by using colored syringe, so that the doctor transfusing the sample, will not be able to know the nature of the sample. From all patients, a right atrial biopsy will be collected for assessment of autologous cardiac stem cells. Also sample of pericardial fluid will be collected for measures of growth factors.

Comparisons: Preoperatively, patients will be imagined by cardiac ultrasound, cardiac MRI, cardiac PET and SPECT. Serum pro-BNB samples will be collected. Postoperatively at 3 months and 6 months pro-BNB and cardiac ultrasound will be evaluated. At one year cardiac ultrasound, cardiac MRI, cardiac PET and SPECT will be reassessed.

Heart failure and coronary artery disease treatments beside the transplantation will be optimized according to the judgment of the doctors of the outpatients clinic. Primary endpoint of the study is the change of ejection fraction in MRI images.

ELIGIBILITY:
Inclusion Criteria:

* General (patients must have all)

  * Symptomatic heart failure.
  * Scheduled to CABG
  * Be 18 to 75 years of age
  * Informed Consent obtained
* Heart Failure Presentation

  * Patients of either gender, who has evaluated in cardiovascular laboratory and scheduled to CABG with moderate heart failure, will be eligible
  * NYHA II-IV symptoms
  * Left ventricular ejection fraction in screening echocardiography 15 to 45%.
  * Optimal heart failure medication and coronary medication before operation, containing at least two heart failure drugs: must have ACE-inhibitor, or AT II blocker, and/or b-blocker together with diuretics, digitalis or aldosterone antagonist, and coronary medication: a statin and anticoagulation, either aspirin or clopidogrel.

Exclusion Criteria:

* Heart failure due to left ventricular outflow track obstruction (valve problem or HOCM)
* History of life-threatening ventricular arrhythmias or resuscitation, condition which may be repeatable or implanted ICD.
* Stroke or other disabling condition with in 3 months before screening
* Contraindications to coronary angiogram or MRI
* Other serious disease limiting life expectancy
* Participation in an other clinical trial
* Severe valve disease: mitral, aortic, tricuspid or pulmonic stenosis / insufficiency
* Scheduled valve operation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2006-10; Primary Completion 2009-12 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
Does a bone marrow transplantation therapy increase the ejection fraction of the heart measured with MRI, when compared with placebo treatment? | 1 year after the transplantation

SECONDARY OUTCOMES:
Does a bone marrow transplantation therapy increase any cardiac function parameter measured by a an echocardiography, MRI or PET ischemia area, when compared with no treatment group? | 6 months and 1 year after the procedure
Does a bone marrow transplantation therapy improve BNP-value? | 3kk, 6 months and 1 year after the procedure
Does a bone marrow transplantation therapy decrease hospitalization or the days stayed in hospital? | primary hospital stay after the transplantation
Does pericardial fluid growth factor concentrations correlate to left ventricular function improvement? | up to 1 year after the translantation
Does autologous cardiac stem cell quality correlate to left ventricular function improvement? | 3kk, 6 months and 1 year after the transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Ari Harjula, MD; PhD, Principal Investigator — Department of Cardiothoracic Surgery, Helsinki University MeilahtiHospital
Locations (1):
- Department of Cardiothoracic Surgery, Meilahti Hospital, Helsinki, Finland

REFERENCES:
- [Derived] Lehtinen M, Patila T, Vento A, Kankuri E, Suojaranta-Ylinen R, Poyhia R, Harjula A; Helsinki BMMC Collaboration. Prospective, randomized, double-blinded trial of bone marrow cell transplantation combined with coronary surgery - perioperative safety study. Interact Cardiovasc Thorac Surg. 2014 Dec;19(6):990-6. doi: 10.1093/icvts/ivu265. Epub 2014 Aug 20. PMID 25142068
- [Derived] Patila T, Lehtinen M, Vento A, Schildt J, Sinisalo J, Laine M, Hammainen P, Nihtinen A, Alitalo R, Nikkinen P, Ahonen A, Holmstrom M, Lauerma K, Poyhia R, Kupari M, Kankuri E, Harjula A. Autologous bone marrow mononuclear cell transplantation in ischemic heart failure: a prospective, controlled, randomized, double-blind study of cell transplantation combined with coronary bypass. J Heart Lung Transplant. 2014 Jun;33(6):567-74. doi: 10.1016/j.healun.2014.02.009. Epub 2014 Feb 14. PMID 24656645